CLINICAL TRIAL: NCT05539794
Title: Exercise Intervention for Adolescents With Cancer (EXERCADOL): A Randomized Controlled Trial
Brief Title: Exercise in Adolescents With Cancer (EXERCADOL)
Acronym: EXERCADOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad Europea de Madrid
Record Dates: First submitted 2022-04-18; First posted 2022-09-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Cancer
Keywords: cancer; lifestyle; cardiac function
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The investigators will apply a two-arm RCT design, following the Consolidated Standards of Reporting Trials recommendations (1:1 randomisation ratio using a computer-generated random allocation sequence with a block on sex and main tumour type [leukaemias/solid tumours]).
Who Masked: Outcomes Assessor
Masking Description: Assessment staff will be blinded to participant randomisation assignment. Yet, because of the nature of the study, it will not be possible to conceal the group assignment from the staff (i.e., fitness specialists) involved in the intervention (physical exercise) sessions. Participants will be explicitly informed on the group to which they will be assigned as well as on the study hypotheses and will be reminded not to discuss their randomisation assignments with assessment staff and/or other patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will follow a supervised physical exercise program.
  Interventions: Behavioral: Physical exercise
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Physical exercise — the intervention group will follow a supervised physical exercise intervention--see below.
  The exercise program (3 supervised sessions/week of aerobic and muscle strength exercises) will be performed: (a) in the hospital gymnasium, or (b) in the patients' room (during phases of treatment-induced immunodepression, where isolation is needed to prevent infections), or (c) online (for those unable to attend the hospital on that day/s). It will also include specific training of the respiratory ('inspiratory') muscles (e.g., diaphragm) on 5 days/week.
  Arms: Intervention

SUMMARY:
The investigators will study the effects of an supevised exercise intervention along the duration of intensive treatment (neoadjuvant [solid tumours]/intense chemotherapy [leukemias], expected median duration 5-6 months) on several health-related variables. Participants will be recruited from 4 hospitals in Madrid (Spain). Inclusion criteria: male/female aged 12-19 years, newly diagnosed--or relapse of-- a malignant extracranial tumour; not having received any type of therapy--except surgery--at the time of diagnosis; adequate health status (Karnofsky/Eastern Cooperative Oncology Group scale score ≥50/≤2); to understand Spanish language and to provide written informed consent. The investigators will recruit ≥136 participants and conduct a randomised controlled trial. The intervention group will follow a supervised concurrent exercise program from the start to the end of intensive treatment. The exercise intervention will be performed in the hospital gymnasium or in the patients' ward (during neutropenic phases), and will also include supervised online sessions. Additionally, the intervention group will perform include inspiratory muscle training. The following outcomes will be assessed at baseline (diagnosis), end of treatment, and at 3-month follow-up in all participants: echocardiography-determined left ventricular function (primary outcome); and other echocardiography-determined variables, cardiac biomarkers, blood pressure, blood lipids, body composition, physical activity levels, energy intake, cardiorespiratory fitness, muscle strength, functional mobility, health-related quality of life, cancer-related fatigue, clinical variables, and potential biological underpinnings of exercise multisystemic benefits (metabolic and inflammatory markers, plasma proteome, gut microbiome, and immune function).

DETAILED DESCRIPTION:
Background. Health promotion interventions are needed during adolescent cancer treatment to facilitate the acquisition of good health practices as patients transition to survivorship. Although meta-analytical evidence supports the health benefits of exercise in the context of childhood cancer, there is scant data focusing solely on adolescents.

Hypothesis and objectives. The investigators hypothesise that a supervised exercise intervention combined with lifestyle counselling during treatment for adolescent cancer will provide several health benefits, particularly related to the cardiometabolic profile. Thus, the investigators will study the effects of a supervised exercise intervention along the duration of intensive treatment (neoadjuvant [solid tumours]/intense chemotherapy [leukaemias], expected median duration 5-6 months) on several health-related variables.

Setting and Methods. Participants will be recruited from 4 hospitals in Madrid (Spain). Inclusion criteria: male/female aged 12-19 years, newly diagnosed with (or having relapse of) a malignant extracranial tumour; not having received any type of therapy--except surgery--at the time of diagnosis; adequate health status (Karnofsky/Eastern Cooperative Oncology Group scale score ≥50/≤2); to understand Spanish language and to provide written informed consent. The investigators will recruit ≥136 participants and conduct a randomised controlled trial (1:1 ratio randomisation with a block on gender and tumour type [leukaemias/lymphomas]). In addition to usual care, the two groups will receive health counselling twice a month (i.e., psychological intervention based on motivational interviewing techniques, as well as guidance on heathy activity, sleeping, and dietary habits). The intervention group will follow a physical exercise and lifestyle counselling program. The exercise intervention will be performed in the hospital gymnasium (3 sessions/week of aerobic and resistance exercises), except for neutropenic phases--during which time sessions will be performed in the patients' ward--and will also include online sessions. Inspiratory muscle training (5 days/week) will be also performed. Patients in the control group will have the option to go to the hospital gymnasium twice a month (to perform playing activities) in order to maximize compliance to the study and to maintain contact with them. The following outcomes will be assessed at baseline (diagnosis), end of treatment, and at 3-month follow-up in all participants: echocardiography-determined left ventricular function (primary outcome); and other echocardiographic variables, cardiometabolic biomarkers, blood pressure, blood lipids, dual-energy X-ray absorptiometry-determined body composition (fat [including visceral adipose tissue]/lean mass, bone mineral content/density), energy intake, cardiorespiratory fitness, muscle strength, functional mobility, health-related quality of life, cancer-related fatigue, clinical variables (survival, treatment tolerability, hospitalisation length), and potential biological underpinnings of exercise multisystemic benefits (cardiometabolic and inflammatory biomarkers, gut microbiome, and immune function [lymphocyte subpopulations, natural killer cell cytotoxicity]) (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with a malignant extracranial tumour
* Not having received any therapy--except surgery--at diagnosis
* Adequate health status (Karnofsky/Eastern Cooperative Oncology Group scale score ≥50/2)
* To understand Spanish language and provide written informed consent.

Exclusion Criteria:

* Life expectancy <3 months
* Comorbidity/acute condition contraindicating exercise practice

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in left-ventricular (LV) function (LV ejection fraction) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined LV ejection fraction (unit = %)
Change in left-ventricular (LV) function (LV ejection fraction) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Echocardiography-determined LV ejection fraction (unit = %)
Change in left-ventricular (LV) function (LV fractional shortening) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined LV fractional shortening (unit = %)
Change in left-ventricular (LV) function (LV fractional shortening) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)]
  Echocardiography-determined LV fractional shortening (unit = %)
Change in global longitudinal strain (GLS) of the left ventricle from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined GLS (%)
Change in global longitudinal strain (GLS) of the left ventricle from baseline to 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Echocardiography-determined GLS (%)

SECONDARY OUTCOMES:
Change in 'clinic' arterial blood pressure from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis
  Arterial blood pressure (BP) (units = mmHg)
Change in 'clinic' arterial blood pressure from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Arterial blood pressure (BP) (units = mmHg)
Change in serum lipid profile (cholesterol) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis)]
  Total/HDL/LDL-cholesterol will be quantified with an automated chemistry analyser (units = mg/dL).
Change in serum lipid profile (cholesterol) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)]
  Total/HDL/LDL-cholesterol will be quantified with an automated chemistry analyser (units = mg/dL).
Change in serum lipid profile (triglycerides) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis)]
  Tiglycerides will be quantified with an automated chemistry analyser (units = mg/dL).
Change in serum lipid profile (triglycerides) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)]
  Tiglycerides will be quantified with an automated chemistry analyser (units = mg/dL).
Change in adiposity index from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Waist-to-hip ratio (no units)
Change in adiposity index from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); (2) 3 months after the end of treatment (follow-up)
  Waist-to-hip ratio (no units)
Change in DXA measures of lean mass from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  DXA-determined total lean mass (grams)
Change in DXA measures of lean mass from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  DXA-determined total lean mass (grams)
Change in DXA measures of fat mass from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  DXA-determined total fat mass (grams)
Change in DXA measures of fat mass from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  DXA-determined total fat mass (grams)
Change in DXA measure of bone mineral density of the total body (less head) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  DXA-determined subtotal bone mineral density (unit = g/cm2)
Change in DXA measure of bone mineral density of the total body (less head) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and 3 months after the end of treatment (follow-up)
  DXA-determined subtotal bone mineral density (unit = g/cm2)
Change in cardiorespiratory fitness (VO2peak) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  VO2peak will be determined with 'breath-by breath' analysis of expired gases on a metabolic cart using a ramp-like bicycle- or arm-crank ergometer -for those participants missing a lower limb- test (units = mL/kg/min)
Change in cardiorespiratory fitness (VO2peak) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  VO2peak will be determined with 'breath-by breath' analysis of expired gases on a metabolic cart using a ramp-like bicycle- or arm-crank -for those participants missing a lower limb- ergometer test (units = mL/kg/min).
Change in muscle strength from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  The 5-repetition maximum (commonly abbreviated as 5RM), which is the maximum strength capacity to perform 5 repetitions until momentary muscular exhaustion, will be measured for leg press and bench press, as well as for seated lateral row, lateral pull down and knee extension (units = kg).
Change in muscle strength from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis);and (2) 3 months after the end of treatment (follow-up)
  The 5-repetition maximum (commonly abbreviated as 5RM), which is the maximum strength capacity to perform 5 repetitions until momentary muscular exhaustion, will be measured for leg press and bench press, as well as for seatead lateral row, lateral pull down and knee extension (units = kg).
Change in inspiratory muscle strength (PImax) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  PImax (units = cmH20) will be determined using a mouth pressure meter with the best result from 3 attempts (interspersed with rest periods of ≥1 min-duration) taken.
Change in inspiratory muscle strength (PImax) from baseline to follow-up | Assessed at three time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  PImax (units = cmH20) will be determined using a mouth pressure meter with the best result from 3 attempts (interspersed with rest periods of ≥1 min-duration) taken.
Survival from baseline to follow-up | Assessed from baseline (diagnosis) until 3 months after end of treatment (follow-up)
  Number of days elapsed from diagnosis until the end of the study (or death, tumor recurrence, or transplant)
Treatment tolerability from baseline to end of treatment | Assessed from baseline (diagnosis) until 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Number of days of treatment interruption/delay
Change in clinical variables (days of hospitalization) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis
  Total hospitalisation length (number of days)
Change in clinical variables (global score of Common Terminology Criteria for Adverse Events [CTCAE]) from baseline to end of treatment | Assessed continuously (every day) from baseline (diagnosis) until 14 to 28 weeks after diagnosis.
  Common Terminology Criteria for Adverse Events [CTCAE, global score, 1 (low toxicity) to 5 (highest)]
Change in clinical variables (global score of Common Terminology Criteria for Adverse Events [CTCAE]) from baseline to follow-up | Assessed continuously (every day) from baseline (diagnosis) until 3 months after the end of treatment (follow-up)
  Common Terminology Criteria for Adverse Events [CTCAE, global score, 1 (low toxicity) to 5 (highest])
Change in metabolic markers (glucose) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis
  Serum fasting glycaemia (mg/dL)
Change in metabolic markers (glucose) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Serum fasting glycaemia (mg/dL)
Change in metabolic markers (insulin) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Serum fasting insulinaemia (pmol/L)
Change in metabolic markers (insulin) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Serum fasting insulinaemia (pmol/L)
Change in metabolic markers (HOMA-IR) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Homeostasis model assessment-insulin resistance index (HOMA-IR) (molar units)
Change in metabolic markers (HOMA-IR) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Homeostasis model assessment-insulin resistance index (HOMA-IR) (molar units)
Change in chronic systemic inflammation (high-sensitivity C-reactive protein) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  High-sensitivity C-reactive protein (mg/L)
Change in chronic systemic inflammation (high-sensitivity C-reactive protein) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  High-sensitivity C-reactive protein (mg/L)
Change in plasma cardiometabolic-related targeted proteome from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Olink® cardiometabolic reagent kit, which measures 92 cardiometabolic related human protein biomarkers simultaneously (units = Normalized Protein Expression (NPX) values, Olink's arbitrary unit presented in log2 scale)
Change in plasma cardiometabolic-related targeted proteome from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (i.e., follow-up)
  Olink® cardiometabolic reagent kit, which measures 92 cardiometabolic related human protein biomarkers simultaneously (units = Normalized Protein Expression (NPX) values, Olink's arbitrary unit presented in log2 scale)
Change in gut microbiome (alpha-diversity) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  α-diversity
Change in gut microbiome (alpha-diversity) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  α-diversity
Change in gut microbiome (beta-diversity) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  beta-diversity
Change in gut microbiome (beta-diversity) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Beta-diversity
Change in gut microbiome (specific bacteria) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Changes in bacteria abundance
Change in gut microbiome (specific bacteria) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Changes in bacteria abundance
Change in Immune phenotype (lymphocyte subpopulations) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis
  Lymphocyte subpopulations (%)
Change in Immune phenotype (lymphocyte subpopulations) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Lymphocyte subpopulations (%)
Change in Immune phenotype (natural killer (NK) cells) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  NK cell subsets (%)
Change in Immune phenotype (NK cells) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  NK cell subsets (%)
Change in Immune function from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  NK cell receptors
Change in immune function from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  NK cell receptors
Change in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) from baseline to end of treatment | : Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  NT-proBNP (units = pg/mL)
Change in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) from baseline to 3 months after the end of treatment (follow-up) | : Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  NT-proBNP (units = pg/mL)
Change in cardiac troponin I from baseline to end of treatment | : Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Cardiac troponin I (units = ng/mL)
Change in cardiac troponin I from baseline to 3 months after the end of treatment (follow-up) | : Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Cardiac troponin I (units = ng/mL)
Change in left-ventricular (LV) mass from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined LV mass (unit = grams)
Change in left-ventricular (LV) mass from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) and (2) 3 months after the end of treatment (follow-up)
  Echocardiography-determined LV mass (unit = grams)
Change in relative wall thickness (RWT) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined RWT (units = cm)
Change in relative wall thickness (RWT) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Echocardiography-determined RWT (units = cm)
Change in DXA measures of visceral adipose tissue (VAT) from baseline to end of tratment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  DXA-determined VAT (unit = grams)
Change in DXA measures of visceral adipose tissue (VAT) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  DXA-determined VAT (grams)
Change in serum lipid profile (apolipoprotein B) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Apolipoprotein B will be quantified with an automated chemistry analyser (units = mg/dL).
Change in serum lipid profile (apolipoprotein B) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis)]
  Apolipoprotein B will be quantified with an automated chemistry analyser (units = mg/dL).
Change in handgrip strength from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Handgrip strength will be measured in both dominant and non-dominant arm (units = kg).
Change in handgrip strength from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis);and (2) 3 months after the end of treatment (follow-up)
  Handgrip strength will be measured in both dominant and non-dominant arm (units = kg).
Change in interventricular septum thickness (IVS) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined IVS (units = mm)
Change in interventricular septum thickness (IVS) from baseline to 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Echocardiography-determined IVS (mm)
Change in left-ventricular end-diastolic diameter (LVEDD) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined LVEDD (mL)
Change in left-ventricular LV end-diastolic diameter (LVEDD) from baseline to 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Echocardiography-determined LVEDD (mL)
Change in left-ventricular posterior wall thickness (LVPW) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Echocardiography-determined LVPW (mm)
Change in left-ventricular posterior wall thickness (LVPW) from baseline to 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Echocardiography-determined LVPW (mm)
Change in functional mobility (Timed Up and Go (TUG)) test) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Performance in TUG test (seconds)
Change in functional mobility (Timed Up and Go (TUG)) test) from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Performance in TUG test (seconds)
Change in functional mobility (Timed Up and Down Stairs (TUDS)) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Performance in TUDS test (units = seconds)
Change in functional mobility (Timed Up and Down Stairs (TUDS) test) from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Performance in TUDS test (seconds)
Change in functional mobility (30-second chair stand test) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Performance in 30-second chair stand test (unit = number of repetitions)
Change in functional mobility (in 30-second chair stand test) from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Performance in in 30-second chair stand test (units = number of repetitions)
Change in health-related quality of life (HRQoL) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Paediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module (Patient's version), designed to measure paediatric/adolescent cancer specific HRQoL (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in health-related quality of life (HRQoL) from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Paediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module (Patient's version), designed to measure paediatric/adolescent cancer specific HRQoL (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in fatigue from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Cancer-related fatigue (Paediatric Quality of Life (PedsQL)) Multidimensional Fatigue Scale, Patient's version (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in fatigue from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Cancer-related fatigue (Paediatric Quality of Life (PedsQL)) Multidimensional Fatigue Scale, Patient's version (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in energy and nutrient intake from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Energy (total kcal/day) and substrate (carbohydrate, fat, protein, all in grams) intake, as estimated using the Nutrimind software based on the participants' reported food consumption frequencies in questionnaires
Change in energy and nutrient intake from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Energy (total kcal/day) and substrate (carbohydrate, fat, protein, all in grams) intake, as estimated using the Nutrimind software based on the participants' reported food consumption frequencies in questionnaires
Change in body mass index (BMI) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  BMI (weight (kg)/height squared (m2))
Change in body mass index (BMI) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); (2) 3 months after the end of treatment (follow-up)
  BMI (weight (kg)/height squared (m2))
Change in DXA measure of bone mineral density of the femoral neck from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment).
  DXA-determined bone mineral density of the femoral neck (unit = g/cm2)
Change in DXA measure of bone mineral density of the femoral neck from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and 3 months after the end of treatment (follow-up)
  DXA-determined total bone mineral density of the femoral neck (unit = g/cm2)
Change in peak power output (also known was 'peak work capacity') from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Peak power output will be determined using a ramp-like cycle- or crank-ergometer-for those participants missing a lower limb-test (units = watts/kg)
Change in in peak power output (also known was 'peak work capacity') from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Peak power output will be determined using a ramp-like cycle- or crank-ergometer-for those participants missing a lower limb-test (units = watts/kg)
Change in the power output eliciting the 'ventilatory threshold' from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)]
  The ventilatory threshold will be visually determined with 'breath-by breath' analysis of expired gases on a metabolic cart using a ramp-like cycle- or crank-ergometer-for those participants missing a lower limb-test (units = watts/kg)
Change in the power output eliciting the 'ventilatory threshold' from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  The ventilatory threshold will be visually determined with 'breath-by breath' analysis of expired gases on a metabolic cart using a ramp-like cycle- or crank-ergometer-for those participants missing a lower limb-test (units = watts/kg)
Change in health-related quality of life (HRQoL) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Paediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module (Parent's version), designed to measure paediatric/adolescent cancer specific HRQoL (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in health-related quality of life (HRQoL) from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Paediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module (Parent's version), designed to measure paediatric/adolescent cancer specific HRQoL (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in fatigue from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Cancer-related fatigue (Paediatric Quality of Life (PedsQL)) Multidimensional Fatigue Scale, Parent's version (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in fatigue from baseline 3 months after the end of treatment (follow-up) | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Cancer-related fatigue (Paediatric Quality of Life (PedsQL)) Multidimensional Fatigue Scale, Parents' version (0 to 100 scale, with higher scores indicating better HRQoL). Units = 0 to 100.
Change in the range of movement (ROM) of the ankle in the relaxed position from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Ankle's ROM in the relaxed position will be assessed using a goniometer, except for those patients with an amputated ankle or a tumor next to the ankle (units = º)
Change in the range of movement (ROM) of the ankle in the relaxed position from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); (2) 3 months after the end of treatment (follow- up)
  Ankle's ROM in the relaxed position will be assessed using a goniometer, except for those patients with an amputated ankle or a tumor next to the ankle (units = º)
Change in the range of movement (ROM) of the ankle at dorsiflexion from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Ankle's ROM at dorsiflexion will be assessed using a goniometer, except for those patients with an amputated ankle or a tumor next to the ankle (units = º)
Change in the range of movement (ROM) of the ankle at dorsiflexion from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment (follow-up)
  Ankle's ROM at dorsiflexion will be assessed using a goniometer, except for those patients with an amputated ankle or a tumor next to the ankle (units = º)
Change in the physical activity levels from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Physical activity levels will be measured with the 'Youth Activity Profile' (YAP) questionnaire
Change in the physical activity levels from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment
  Physical activity levels will be measured with the 'Youth Activity Profile' (YAP) questionnaire
Change in the physical activity levels from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Physical activity levels will be measured with the 'Assessment of Physical Activity Levels' (APAL) questionnaire (units = score from 5 to 20)
Change in the physical activity levels from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment
  Physical activity levels will be measured with the 'Assessment of Physical Activity Levels' (APAL) questionnaire (units = score from 5 to 20)
Change in the number of viral/bacterial/fungal infections from baseline to end of treatment | Assessed continuously (every day) from baseline (diagnosis) until 14 to 28 weeks after diagnosis (i.e., end of treatment)
  The number of viral/bacterial/fungal infections will be retrieved from medical records
Change in the number of viral/bacterial/fungal infections from baseline to follow-up | Assessed continuously (every day) from baseline (diagnosis) until 3 months after the end of treatment
  The number of viral/bacterial/fungal infections will be retrieved from medical records
Change in metabolic markers (glycated hemoglobin) from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Serum fasting glycated hemoglobin (mmol/mol)
Change in metabolic markers (glycated hemoglobin) from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment
  Serum fasting glycated hemoglobin (mmol/mol)
Change in left-ventricular (LV) hypertrophy from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Age-specific >95th percentile for LV mass
Change in left-ventricular (LV) hypertrophy from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment
  Age-specific >95th percentile for LV mass
Change in VO2 at the ventilatory threshold from baseline to end of treatment | Assessed at two time points: (1) at baseline (diagnosis); and (2) 14 to 28 weeks after diagnosis (i.e., end of treatment)
  VO2 at the ventilatory threshold will be determined with 'breath-by breath' analysis of expired gases on a metabolic cart using a ramp-like bicycle- or arm-crank ergometer -for those participants missing a lower limb- test (units = mL/kg/min)
Change in VO2 at the ventilatory threshold from baseline to follow-up | Assessed at two time points: (1) at baseline (diagnosis); and (2) 3 months after the end of treatment
  VO2 at the ventilatory threshold will be determined with 'breath-by breath' analysis of expired gases on a metabolic cart using a ramp-like bicycle- or arm-crank ergometer -for those participants missing a lower limb- test (units = mL/kg/min)
Change in toxicity grade from baseline to end of treatment | Assessed continuously (every day) from baseline (diagnosis) until 14 to 28 weeks after diagnosis (i.e., end of treatment)
  Toxicity grade will be assessed using the formula from Langlais et al (2022), where using the 5 adverse events of higher grade, provides a score from 5 (more toxicity) to 0 (less toxicity)
Change in toxicity grade from baseline to follow-up | Assessed continuously (every day) from baseline (diagnosis) until 3 months after the end of treatment
  Toxicity grade will be assessed using the formula from Langlais et al (2022), where using the 5 adverse events of higher grade, provides a score from 5 (more toxicity) to 0 (less toxicity)
Change in the duration of viral/bacterial/fungal infections from baseline to end of treatment | Assessed continuously (every day) from baseline (diagnosis) until 14 to 28 weeks after diagnosis (i.e., end of treatment)
  The duration of viral/bacterial/fungal infections will be retrieved from medical records
Change in the duration of viral/bacterial/fungal infections from baseline to follow-up | Assessed continuously (every day) from baseline (diagnosis) until 3 months after the end of treatment
  The duration of viral/bacterial/fungal infections will be retrieved from medical records
Adherence to the exercise intervention from baseline to end of treatment | Assessed continuously (every day) from baseline (diagnosis) until 14 to 28 weeks after diagnosis (i.e., end of treatment)
  The number of attended exercise sessions

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Universidad Europea de Madrid, Villaviciosa de Odón, Spain
  - UEM, Madrid

IPD SHARING:
Plan to Share IPD: No
As per Spanish regulations